CLINICAL TRIAL: NCT06254755
Title: Comparison of Clinical and Radiological Outcomes Between Suction Aspiration Method and Combination Method of Intra-arterial Therapy (IAT) in Large Artery Occlusion: Randomized Open-labelled Prospective Multicenter Trials
Brief Title: Comparison Study Between Suction Aspiration and Combination Technique in Acute Cerebral Infarction
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Inje University Haeundae Paik Hospital (Other)
Collaborators: Korean Neuroendovascular Society (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HaeundaePaikH
Record Dates: First submitted 2024-01-17; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Acute Cerebral Ischemia Requiring for Mechanical Thrombectomy
Keywords: acute cerebral infarction, mechanical thrombectomy, suction aspiration, combination

STUDY DESIGN:
Intervention Model Description: Non-inferiority, open-labelled, randomization, case-controlled prospective multicenter trials
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- suction aspiration group (Experimental): suction aspiration group is based on a large bore catheter for thrombus removal under negative pressure of pump or manual syringe.
  Interventions: Device: mechanical thrombectomy
- combination group (Active Comparator): combination group is based on a stent retrieval with a large bore catheter for thrombus removal under negative pressure of pump or manual syringe.
  Interventions: Device: mechanical thrombectomy

INTERVENTIONS:
Device: mechanical thrombectomy — mechanical thrombectomy of acute ischemic stroke caused by major vessel occlusion of the anterior circulation has become an accepted procedure in the last decade.

SUMMARY:
Mechanical thrombectomy of acute ischemic stroke caused by major vessel occlusion of the anterior circulation has become an accepted procedure in the last decade. Recent IAT modalities have been classified as suction aspiration,stent retrieval and combination modality. The suction aspiration technique is limited by the possibility of breaking the entire thrombus during the IAT. In addition, the stent retrieval technique is also limited because of thrombus migration during stent removal from an acute-angled artery as in the case of a carotid siphon.

According to recent development of suction catheter, investigators expected that suction aspiration will prevent breaking the entire thrombus during the IAT. Investigators will evaluate the radiological and clinical outcome of suction aspiration technique in comparison with combination technique in the large artery occlusion feasible to both suction aspiration and combination technique prospectively in a randomized trial.

DETAILED DESCRIPTION:
*Hospital code for the participant hospitals Bundang Cha Hospital (A) Inje University Haeundae Paik Hospital(I) Samsung Medical Center Sungkyunkwan University (B) Kosin University Gospel Hospital (C) Daegu Good morning Hospital (D) Yeungnam University Medical Center (E) Pohang S hospital(G) Inje University Ilsan Paik Hospital(H) SM christianity Pohang Hospital(L) Choongnam National University Hospital(N) Inha University Hospital(P) Catholic University of Korea Bucheon ST. Mary's Hospital (Q) Catholic University of Korea Uijeongbu ST. Mary's Hospital (R) Catholic University of Korea ST. Vincent's Hospital (S) Ulsan University Hospital (U)

Alphabetic number of each hospital is an each hospital code.

If the patient with acute cerebral infarction will be feasible to suction aspiration and combination technique, the investigator who can enroll the patient should check the order of random table in open chatting board and perform the ordered method after completion of consent for the COMPETE trials.

Each investigator in the hospitals participated in COMPETE trials will write the competetrials spread sheet on google web.

The image files of thrombectomy including pre-thrombectomy and post-thrombectomy will be converted to zip file and send to the independent neurointerventional radiologist on e-mail about 2 ~ 4 times a year. the independent examiner will re-send to the investigator after completion of modified TICI grade in the image files of thrombectomy.

This study should not enroll atherosclerotic tandem occlusion. Other etiologies such as cancer related stroke or dissection should not be enrolled in this study.

Cases of Atherosclerotic steno-occlusion will be included in this study. Rescue treatment such as primary stenting or conventional modality will be performed according to the favored modality of each investigator.

ELIGIBILITY:
Inclusion Criteria:

* interventionist
* minimal experiences of thrombectomy ≥ 50 cases
* successful recanalization (TICI≥2b) of radiological outcome in all cases treated by thrombectomy > 70% Patient inclusion criteria
* age ≥ 18
* acute cerebral infarction with initial NIHSS ≥ 4
* patients with agreement for clinical trials
* detection of large artery occlusion based on CT or Magnetic resonance angiography
* definition of large artery occlusion: 1) anterior circulation internal carotid artery(ICA), M1, M2 segment A1, A2 segment 2)posterior circulation Vertebrobasilar occlusion including P1 segment
* Last normal time ≤ 24 hours
* Flow/volume mismatch ≥ 1/2 based on perfusion image

Exclusion Criteria:

* Previous disabled patients before mechanical thrombectomy(MT) (Karnofsky performance Status Scale(KPS) ≤ 80)
* Patient or patient's guardian refused to the clinical trial
* Small vessel disease of TOAST classification
* Other determined etiologies of TOAST classification
* Patients with Initial NIHSS ≤ 3
* Diffusion/perfusion matched lesion or flow/volume matched lesion

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1132 (Estimated)
Dates: Start 2022-10-01 (Actual); Primary Completion 2027-01-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Radiological outcome using modified TICI grade (mTICI) | time of control angiography after retrieval of thrombectomy devices
  modified TICI grade is composed of 0, 1, 2a,2b,2c, and 3. O of modified TICI grade is no recanalized state. 3 of modified TICI grade is completely recanalized state.
clinical outcome using modified Rankin Scale(mRS) | 3 months after thrombectomy
  modified Rankin scale is composed of 0,1,2,3,4,5, and. Oof mRS is no neurological deficit. 6 of mRS is mortality case.
Radiological outcome caused by cardioembolism using using modified TICI grade (mTICI) | time of control angiography after retrieval of thrombectomy devices
  modified TICI grade is composed of 0, 1, 2a,2b,2c, and 3. O of modified TICI grade is no recanalized state. 3 of modified TICI grade is completely recanalized state.
clinical outcome cause by cardioembolism using modified Rankin Scale(mRS) | 3 months after thrombectomy
  modified Rankin scale is composed of 0,1,2,3,4,5, and. Oof mRS is no neurological deficit. 6 of mRS is mortality case.
radiological outcome in M1 occlusion using modified TICI grade (mTICI) | time of control angiography after retrieval of thrombectomy devices
  modified TICI grade is composed of 0, 1, 2a,2b,2c, and 3. O of modified TICI grade is no recanalized state. 3 of modified TICI grade is completely recanalized state.
clinical outcome in M1 occlusion using modified Rankin Scale(mRS) | 3 months after thrombectomy
  modified Rankin scale is composed of 0,1,2,3,4,5, and. Oof mRS is no neurological deficit. 6 of mRS is mortality case.
radiological outcome in M2 occlusion using modified TICI grade (mTICI) | time of control angiography after retrieval of thrombectomy devices
  modified TICI grade is composed of 0, 1, 2a,2b,2c, and 3. O of modified TICI grade is no recanalized state. 3 of modified TICI grade is completely recanalized state.
clinical outcome in M2 occlusion using modified Rankin Scale(mRS) | 3 months after thrombectomy
  modified Rankin scale is composed of 0,1,2,3,4,5, and. Oof mRS is no neurological deficit. 6 of mRS is mortality case.
comparison of clinical outcome 3 months after IAT between mismatch more than 1/2 based on flow/volume of CT perfusion and calculated volume of mismatch using modified Rankin Scale(mRS) | 3 months after thrombectomy
  modified Rankin scale is composed of 0,1,2,3,4,5, and. Oof mRS is no neurological deficit. 6 of mRS is mortality case.
comparison of radiological outcome between more than 1/2 based on flow/volume of CT perfusion and calculated volume of mismatch based on flow/volume of CT perfusion | time of control angiography after retrieval of thrombectomy devices
  modified TICI grade is composed of 0, 1, 2a,2b,2c, and 3. O of modified TICI grade is no recanalized state. 3 of modified TICI grade is completely recanalized state.
comparison of radiological outcome between rescue treatment of primary stenting and sequential treatment in large artery atherosclerotic steno-occlusion using modified TICI grade (mTICI) | time of control angiography after retrieval of thrombectomy devices
  modified TICI grade is composed of 0, 1, 2a,2b,2c, and 3. O of modified TICI grade is no recanalized state. 3 of modified TICI grade is completely recanalized state.
comparison of clinical outcome 3 months after IAT between rescue treatment of primary stenting and sequential treatment in large artery atherosclerotic steno-occlusion using modified Rankin Scale(mRS) | 3 months after thrombectomy
  modified Rankin scale is composed of 0,1,2,3,4,5, and. Oof mRS is no neurological deficit. 6 of mRS is mortality case.
comparison of door-to-puncture time between hot-line prehospital tele-communication and conventional group | time interval from ER arrival time to femoral puncture
  time interval between emergent room arrival time and femoral puncture
comparison of radiological outcome between hot-line prehospital tele-communication and conventional group using modified TICI grade (mTICI) | time of control angiography after retrieval of thrombectomy devices
  modified TICI grade is composed of 0, 1, 2a,2b,2c, and 3. O of modified TICI grade is no recanalized state. 3 of modified TICI grade is completely recanalized state.
comparison of clinical outcome 3 months after IAT between hot-line prehospital tele-communication and conventional group using modified Rankin Scale(mRS) | 3 months after thrombectomy
  modified Rankin scale is composed of 0,1,2,3,4,5, and. Oof mRS is no neurological deficit. 6 of mRS is mortality case.

SECONDARY OUTCOMES:
switching rate | time of switching from combination technique to suction aspiration
  switching rate from combination technique to suction aspiration technique
switching rate | time of switching from suction aspiration to combination technique
  switching rate from suction aspiration technique to combination technique
recanalization failure rate | time of final control angiogram immediately after thrombectomy
  recanalization failure rate of IAT
procedure related complication | admission period
  procedural morbidity and mortality rate
non-procedural morbidity and mortality rate | admission period
  non-procedure related events and death such as myocardial infarction, pneumonia, or sepsis

CONTACTS AND LOCATIONS:
Overall Officials: Sung-Chul Jin, PhD, Principal Investigator — Department of Neurosurgery, Inje University, Haeundae Paik Hospital
Locations (13):
- South Korea (13):
  - Inje University Ilsan Paik Hospital, Goyang-si, Gyeonggi-do
  - Bundang Cha Hospital, Seongnam-si, Gyeonggi-do
  - Samsung Medical Center Sungkyunkwan University, Changwon, Gyeongsangnam-do
  - The Catholic University of Korea, Bucheon ST. Mary's Hospital, Bucheon-si
  - Daegu Goodmorning Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Chungnam National University Hospital., Daejeon
  - Inha University Hospital, Incheon
  - Pohang S hospital, Pohang
  - Pohang SM christianity Hospital, Pohang
  - The Catholic University of Korea ST. Vincent's Hospital., Suwon
  - The Catholic University of Korea Uijeongbu St. Mary's Hospital, Uijeongbu-si
  - Ulsan university Hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goto S, Ohshima T, Ishikawa K, Yamamoto T, Shimato S, Nishizawa T, Kato K. A Stent-Retrieving into an Aspiration Catheter with Proximal Balloon (ASAP) Technique: A Technique of Mechanical Thrombectomy. World Neurosurg. 2018 Jan;109:e468-e475. doi: 10.1016/j.wneu.2017.10.004. Epub 2017 Oct 13. PMID 29038080
- [Background] Massari F, Henninger N, Lozano JD, Patel A, Kuhn AL, Howk M, Perras M, Brooks C, Gounis MJ, Kan P, Wakhloo AK, Puri AS. ARTS (Aspiration-Retriever Technique for Stroke): Initial clinical experience. Interv Neuroradiol. 2016 Jun;22(3):325-32. doi: 10.1177/1591019916632369. Epub 2016 Feb 22. PMID 26908591
- [Background] Maegerlein C, Monch S, Boeckh-Behrens T, Lehm M, Hedderich DM, Berndt MT, Wunderlich S, Zimmer C, Kaesmacher J, Friedrich B. PROTECT: PRoximal balloon Occlusion TogEther with direCt Thrombus aspiration during stent retriever thrombectomy - evaluation of a double embolic protection approach in endovascular stroke treatment. J Neurointerv Surg. 2018 Aug;10(8):751-755. doi: 10.1136/neurintsurg-2017-013558. Epub 2017 Dec 8. PMID 29222393
- [Background] Lee DH, Sung JH, Kim SU, Yi HJ, Hong JT, Lee SW. Effective use of balloon guide catheters in reducing incidence of mechanical thrombectomy related distal embolization. Acta Neurochir (Wien). 2017 Sep;159(9):1671-1677. doi: 10.1007/s00701-017-3256-3. Epub 2017 Jul 9. PMID 28691137
- [Background] Brinjikji W, Starke RM, Murad MH, Fiorella D, Pereira VM, Goyal M, Kallmes DF. Impact of balloon guide catheter on technical and clinical outcomes: a systematic review and meta-analysis. J Neurointerv Surg. 2018 Apr;10(4):335-339. doi: 10.1136/neurintsurg-2017-013179. Epub 2017 Jul 28. PMID 28754806
- [Background] Karanam LSP, Sharma M, Alurkar A, Baddam SR, Pamidimukkala V, Polavarapu R. Balloon Angioplasty for Intracranial Atherosclerotic Disease: A Multicenter Study. J Vasc Interv Neurol. 2017 Jun;9(4):29-34. PMID 28702117
- [Result] Maegerlein C, Berndt MT, Monch S, Kreiser K, Boeckh-Behrens T, Lehm M, Wunderlich S, Zimmer C, Friedrich B. Further Development of Combined Techniques Using Stent Retrievers, Aspiration Catheters and BGC : The PROTECTPLUS Technique. Clin Neuroradiol. 2020 Mar;30(1):59-65. doi: 10.1007/s00062-018-0742-9. Epub 2018 Nov 9. PMID 30413831
- [Result] Malisch TW, Zaidat OO, Castonguay AC, Marden FA, Gupta R, Sun CJ, Martin CO, Holloway WE, Mueller-Kronast N, English J, Linfante I, Dabus G, Bozorgchami H, Xavier A, Rai AT, Froehler M, Badruddin A, Nguyen TN, Taqi MA, Abraham MG, Janardhan V, Shaltoni H, Novakovic R, Yoo AJ, Abou-Chebl A, Chen PR, Britz GW, Kaushal R, Nanda A, Nogueira RG. Clinical and Angiographic Outcomes with the Combined Local Aspiration and Retriever in the North American Solitaire Stent-Retriever Acute Stroke (NASA) Registry. Interv Neurol. 2018 Feb;7(1-2):26-35. doi: 10.1159/000480353. Epub 2017 Oct 11. PMID 29628942
- [Result] Maegerlein C, Prothmann S, Lucia KE, Zimmer C, Friedrich B, Kaesmacher J. Intraprocedural Thrombus Fragmentation During Interventional Stroke Treatment: A Comparison of Direct Thrombus Aspiration and Stent Retriever Thrombectomy. Cardiovasc Intervent Radiol. 2017 Jul;40(7):987-993. doi: 10.1007/s00270-017-1614-4. Epub 2017 Mar 7. PMID 28271328
- [Result] Lapergue B, Blanc R, Costalat V, Desal H, Saleme S, Spelle L, Marnat G, Shotar E, Eugene F, Mazighi M, Houdart E, Consoli A, Rodesch G, Bourcier R, Bracard S, Duhamel A, Ben Maacha M, Lopez D, Renaud N, Labreuche J, Gory B, Piotin M; ASTER2 Trial Investigators. Effect of Thrombectomy With Combined Contact Aspiration and Stent Retriever vs Stent Retriever Alone on Revascularization in Patients With Acute Ischemic Stroke and Large Vessel Occlusion: The ASTER2 Randomized Clinical Trial. JAMA. 2021 Sep 28;326(12):1158-1169. doi: 10.1001/jama.2021.13827. PMID 34581737
- [Result] Delgado Almandoz JE, Kayan Y, Young ML, Fease JL, Scholz JM, Milner AM, Hehr TH, Roohani P, Mulder M, Tarrel RM. Comparison of clinical outcomes in patients with acute ischemic strokes treated with mechanical thrombectomy using either Solumbra or ADAPT techniques. J Neurointerv Surg. 2016 Nov;8(11):1123-1128. doi: 10.1136/neurintsurg-2015-012122. Epub 2015 Dec 14. PMID 26667250
- [Result] Kim SH, Lee H, Kim SB, Kim ST, Baek JW, Heo YJ, Jeong HW, Kim HJ, Park JH, Kim JS, Jin SC. Hybrid mechanical thrombectomy for acute ischemic stroke using an intermediate aspiration catheter and Trevo stent simultaneously. J Clin Neurosci. 2020 Jun;76:9-14. doi: 10.1016/j.jocn.2020.04.079. Epub 2020 Apr 21. PMID 32327379
- Available data/document: Individual Participant Data Set — http://competetrials@gmail.com